CLINICAL TRIAL: NCT03755297
Title: Effect of the Inhibitors of the Way JAK-STAT on Regulatory B Cells in the Rheumatoid Arthritis
Brief Title: Effect of the Inhibitors of the Way JAK-STAT on Regulatory B Cells
Acronym: JAK-INH2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Default of recruitment
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL17_0393; 2017-A03095-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-26; First posted 2018-11-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Regulatory B cells; JAK/STAT inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rheumatoid arthritis (Other): Patients responding to ACR/EULAR 2010 criteria and Blood sample analysis of patients treated as standard care
  Interventions: Other: Blood sample analysis of patients treated as standard care
- Osteoarthritis (Other): Control patients and Blood sample analysis of patients treated as standard care
  Interventions: Other: Blood sample analysis of patients treated as standard care
- Rheumatoid arthritis with JAK/STAT inhibitors (Other): Standard use of JAK/STAT inhibitors and Blood sample analysis of patients treated as standard care
  Interventions: Other: Blood sample analysis of patients treated as standard care

INTERVENTIONS:
Other: Blood sample analysis of patients treated as standard care — Blood sample to analyse percentage of blood cells (regulatory B cells et T cells)

SUMMARY:
This study will investigate whether inhibitors of the JAK / STAT signaling pathway can increase anti-inflammatory functions of B cells in patients with RA using in vitro and in vivo experiments.

DETAILED DESCRIPTION:
This study will first analyze the effect of inhibitors of the JAK / STAT pathway in vitro on B-cell phenotypes and functions in 30 RA patients and 30 patients with osteoarthritis. It will also study the phenotypes and functions of B cells in RA patients for whom JAK / STAT inhibitor treatment has been prescribed by the patient's usual rheumatologist. The analysis will be done before the start of treatment and 3 months later. The phenotypes of B-cells will be assessed by flow cytometry with intra- and extra-cellular stainings. The functions of B cells will be assessed by their ability to differenciate naïve T cells in coculture.

ELIGIBILITY:
Inclusion criteria:

* General criteria
* Patient, of 18 and more years old
* Subject affiliated to a social security system
* Subject not being in period of exclusion with regard to another protocol
* Absence of pregnancy in the inclusion (date of the last period, use of a contraceptive method, ß -HCG impulsive person in case of doubt)
* Informed consent
* Criteria of inclusion of the group rheumatoid arthritis (in vitro studies):
* Rheumatoid arthritis, corresponding to the the classification ACR / EULAR 2010 criteria
* Criteria of inclusion of the group arthritis (in vitro studies):
* Spinal degenerative osteoarthritis or degenerative osteoarthritis of the members, according to the clinical and radiological elements.
* Criteria of inclusion of the group rheumatoid arthritis, longitudinal study at the patients treated by JAK / STAT inhibitors :
* Rheumatoid Polyarthritis, corresponding to the classification ACR / EULAR 2010 criteria
* Patient to whom a treatment by inhibitor of the way JAK / STAT was proposed in current care of rheumatoid arthritis.

Exclusion criteria:

* General criteria
* Corticosteroid therapy superior to 10 mg / j
* Drip of corticoids in the previous month
* Pregnant or breast-feeding Patients
* Patient under protection(saving) of justice
* Under guardianship Patient or guardianship
* Current Infection
* Criteria of non-inclusion of the group rheumatoid polyarthritis ( in vitro studies):
* Treatment by immunomodulateur or biotherapics (anti-TNF alpha, tocilizumab, abatacept or rituximab) in the previous year
* Criteria of non-inclusion of the group arthritis ( in vitro studies):
* History of autoimmune disease or néoplasie
* Treatment by immunomodulateur or biotherapics (anti-TNF alpha, tocilizumab, abatacept or rituximab)
* Criteria of non-inclusion of the group rheumatoid arthritis, longitudinal study at the patients treated by JAK / STAT inhibitors :

Treatment by rituximab in the previous year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Percentage of regulatory B cells induced by JAKi in vitro | 4 months
  IL-10+ CD19+ cells after in vitro exposure of JAKi

SECONDARY OUTCOMES:
Percentage of regulatory T cells induced by JAKi treated B cells in vitro | 4 months
  CD25hiCD126lo/-CD4+ after 3 days of coculture with JAKi pretreated B cells
Percentage of Th1 induced by JAKi treated B cells in vitro | 4 months
  Interferon gamma+CD4+ after 3 days of coculture with JAKi pretreated B cells

CONTACTS AND LOCATIONS:
Overall Officials: Claire DAIEN, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No